CLINICAL TRIAL: NCT02160626
Title: A Randomized, Double-Blind, Vehicle Controlled, Parallel Group Study of the Dose-Response Profile of A-101 Topical Solution in Subjects With Seborrheic Keratosis.
Brief Title: Dose-Response Profile of A-101 in Subjects With Seborrheic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-202
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Seborrheic Keratosis
Keywords: Seborrheic keratosis; A101
MeSH Terms: conditions — Keratosis, Seborrheic | interventions — N-phenylacetoaminomethylene-DL-p-nitrophenylalanine; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A-101 Vehicle (Placebo Comparator): A-101 Vehicle (placebo) Topical Solution
  Interventions: Drug: A-101 Vehicle
- A-101 (40) Topical Solution (Active Comparator): A-101 (40) Topical Solution - high dose
  Interventions: Drug: A-101 (40) Topical Solution
- A-101 (32.5) Topical Solution (Active Comparator): A-101 (32.5) Topical Solution - low dose
  Interventions: Drug: A-101 (32.5) Topical Solution

INTERVENTIONS:
Drug: A-101 Vehicle — Placebo control
  Arms: A-101 Vehicle
Drug: A-101 (40) Topical Solution — A-101 (40) Topical Solution - high dose
  Arms: A-101 (40) Topical Solution
Drug: A-101 (32.5) Topical Solution — A-101 (32.5) Topical Solution - low dose
  Arms: A-101 (32.5) Topical Solution

SUMMARY:
The main objective of this study is to evaluate the dose-response relationship of two concentrations of A-101 solution when applied to individual seborrheic keratosis (SK) lesions (target lesions) compared with a matching A-101 Solution Vehicle.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the dose-response relationship of two concentrations of A-101solution when applied to individual seborrheic keratosis (SK) lesions (target lesions) compared with a matching A-101 Solution Vehicle.

Each subject will have 4 target lesions on the trunk/extremities.

A further objective is to evaluate the safety and efficacy of two concentrations of A-101 solution and its matching vehicle when applied to SK target lesions on the trunk/extremities.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject has a clinical diagnosis of stable clinically typical seborrheic keratosis
3. Subject has 4 appropriate seborrheic keratosis target lesions, as defined below, on the trunk/extremities:

   * Have a clinically typical appearance
   * Be treatment naïve
   * Have a Physician Lesion Assessment (PLA) of ≥2
   * Have a longest axis that is ≥7mm and ≤15mm
   * Have a longest dimension perpendicular to the longest axis that is ≥7mm and ≤15mm
   * Have a thickness that is ≤2mm
   * Be a discrete lesion
   * Be, when centered in the area outlined by the provided 3cm diameter circular template, the only seborrheic keratosis lesion present
   * Not be in an intertriginous fold
   * Not be in an area where clothing, such as a bra, might cause physical irritation
   * Not be pedunculated.
4. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an active form of birth control for the duration of the study
5. Subject is non-pregnant and non-lactating
6. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of any target lesion or which exposes the subject to an unacceptable risk by study participation
7. Subject is willing and able to follow all study instructions and to attend all study visits
8. Subject is able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. Subject has clinically atypical and/or rapidly growing seborrheic keratosis lesions
2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Leser-Trelat)
3. Subject has a current systemic malignancy
4. Subject has a history of keloid formation or hypertrophic scarring
5. Subject has used any of the following systemic therapies within the specified period prior to Visit 1:

   * Retinoids; 180 days
   * Glucocorticosteroids; 28 days
   * Anti-metabolites (e.g., methotrexate); 28 days
6. Subject has used any of the following topical therapies within the specified period prior to Visit 1 on, or in a proximity to the target lesion, that in the investigator's opinion, interferes with the application of the study medication or the study assessments:

   * LASER, light (e.g., intense pulsed light (IPL), photo-dynamic therapy (PDT)) or other energy based therapy; 180 days
   * Retinoids; 90 days
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-fluorouracil, or ingenol mebutate; 60 days
   * Glucocorticosteroids or antibiotics; 14 days
   * Moisturizers/emollients, sunscreens; 12 hours
7. Subject currently has or has had any of the following within the specified period prior to Visit 1 on or in a proximity to the target lesion that, in the investigator's opinion, interferes with the application of the study medication or the study assessments:

   * A cutaneous malignancy; 180 days
   * Experienced a sunburn; 28 days
   * A pre-malignancy (e.g., actinic keratosis); currently
   * Body art (e.g., tattoos, piercing, etc.); currently
   * Excessive tan; currently
8. Subject has a history of sensitivity to any of the ingredients in the study medications
9. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
10. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Weiss, MD, Principal Investigator — Gwinnett Clinical Research Center, Inc.; Janet Dubois, MD, Principal Investigator — Derm Research, PLLC; David C Wilson, MD, Principal Investigator — The Education & Research Foundation, Inc.; Daniel M Stewart, DO, Principal Investigator — Michigan Center for Research Corp.; Andrew Blauvelt, MD, MBA, Principal Investigator — Oregon Medical Research Center
Locations (5):
- United States (5):
  - Gwinnett Clinical Research Center, Inc., Snellville, Georgia
  - Michigan Center for Research Corp., Clinton Township, Michigan
  - Oregon Medical Research Center, Portland, Oregon
  - DermReseach, Inc., Austin, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 (40%) Topical Solution: A-101 (40%) Topical Solution - high dose
  A-101 (40) Topical Solution: A-101 (40) Topical Solution - high dose
- A-101 (32.5%) Topical Solution: A-101 (32.5%) Topical Solution - low dose
  A-101 (32.5) Topical Solution: A-101 (32.5) Topical Solution - low dose
Period: Overall Study
Arm/Group | A-101 Vehicle | A-101 (40%) Topical Solution | A-101 (32.5%) Topical Solution
Started | 58 | 57 | 57
Completed | 57 | 56 | 56
Not Completed | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Schedule not conducive to study visits | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- A-101 (40%) Topical Solution: A-101 (40%) Topical Solution - high dose
  A-101 (40%) Topical Solution: A-101 (40%) Topical Solution - high dose
- A-101 (32.5%) Topical Solution: A-101 (32.5%) Topical Solution - low dose
  A-101 (32.5%) Topical Solution: A-101 (32.5%) Topical Solution - low dose
- Total: Total of all reporting groups
Arm/Group | A-101 Vehicle | A-101 (40%) Topical Solution | A-101 (32.5%) Topical Solution | Total
Number analyzed (Participants) | 58 | 57 | 57 | 172
Age, Customized [Count of Participants; unit: Participants]
  18-55 | 0 | 0 | 0 | 0
  56-70 | 2 | 1 | 0 | 3
  71 + | 56 | 56 | 57 | 169
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 28 | 91
  Male | 28 | 24 | 29 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 57 | 57 | 57 | 171
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 58 | 56 | 57 | 171
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 57 | 57 | 172
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a six point scale that evaluates the skin coloration of the patient with one being the lightest and 6 being the darkest skin coloration.
  Participants
    1 | 4 | 4 | 3 | 11
    2 | 13 | 27 | 24 | 64
    3 | 30 | 19 | 20 | 69
    4 | 11 | 6 | 10 | 27
    5 | 0 | 1 | 0 | 1
    6 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Per Subject Percentage Target Lesions Judged Clear by the Physician's Lesion Assessment (PLA)
Description: Mean of per-subject percentages of target lesions judged to be clear on the PLA (PLA = 0) at end of study (Visit 8). The PLA is a four point scale from 0 being clear to 3 being most severe lesion.
Time Frame: Baseline, visit 8
Population: Overall number of participants = number of participants completing the study per protocol.
Measure: Mean (Standard Deviation); unit: percentage of lesions cleared
Units Other Than Participants: Lesions
Arm/Group | A-101 Vehicle | A-101 (32.5%) Topical Solution | A-101 (40%) Topical Solution
Number analyzed (Participants) | 57 | 56 | 56
Number analyzed (Lesions) | 228 | 224 | 224
percentage of lesions cleared | 4.82 (15.26) | 26.79 (38.10) | 45.09 (37.06)
Statistical Analysis 1: Comparison: A-101 Vehicle vs A-101 (32.5%) Topical Solution; Test type: Other; p = 0.0003, ANOVA
Statistical Analysis 2: Comparison: A-101 Vehicle vs A-101 (40%) Topical Solution; Test type: Other; p = .0001, ANOVA

2. Secondary Outcome: Mean Change From Baseline to Visit 8 in the Physician's Lesion Assessment
Description: Change from baseline PLA will be calculated for each lesion first, then per-subject mean changes from baseline will be calculated.
  The PLA is a score on a four scale from 0 to 3 with 0 being clear and 3 being the most severe, a lower score indicating a better result. For the mean change in this score, a larger mean change is a better result.
Time Frame: Baseline, visit 8
Population: N = number of participants completing the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Lesions
Arm/Group | A-101 Vehicle | A-101 (32.5%) Topical Solution | A-101 (40%) Topical Solution
Number analyzed (Participants) | 57 | 56 | 56
Number analyzed (Lesions) | 228 | 224 | 224
units on a scale | -0.32 (0.57) | -0.77 (0.67) | -0.91 (0.77)
Statistical Analysis 1: Comparison: A-101 Vehicle vs A-101 (32.5%) Topical Solution; mean change from baseline to Visit 8 PLA will be performed using Analysis of Covariance (ANCOVA) with baseline PLA as the covariate; Test type: Other; p = 0.0001, ANCOVA
Statistical Analysis 2: Comparison: A-101 Vehicle vs A-101 (40%) Topical Solution; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.0001, ANCOVA

3. Secondary Outcome: Proportion of Subjects Who Had at Least 3 of 4 Target Lesions Judged to be Clear on the Physician Lesion Assessment (PLA =0) at Visit 8.
Description: Proportion of Subjects who had at least 3 of 4 target lesions judged to be clear on the Physician Lesion Assessment (PLA =0) at visit 8. The PLA is a 4 point scale evaluating the severity of a lesion with 0 being clear and 3 being the most severe.
Time Frame: Baseline, visit 8
Population: N = number of subjects who completed the study per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Vehicle | A-101 (32.5%) Topical Solution | A-101 (40%) Topical Solution
Number analyzed (Participants) | 57 | 56 | 56
Participants | 0 | 9 | 11
Statistical Analysis 1: Comparison: A-101 Vehicle vs A-101 (32.5%) Topical Solution; Secondary efficacy analyses will also be conducted based on the proportion of subjects who have at least 3 of 4 target lesions judged to be clear on the PLA (PLA=0) at Visit 8. A separate comparison will be made between each active treatment group and the vehicle treatment group using Cochran-Mantel-Haenszel (CMH) tests stratified by site; Test type: Other; p = 0.0016, Cochran-Mantel-Haenszel — For all analyses, two-tail alpha will be set to 0.05 with no adjustment for multiple comparisons; For all analyses, two-tail alpha will be set to 0.05 with no adjustment for multiple comparisons
Statistical Analysis 2: Comparison: A-101 Vehicle vs A-101 (40%) Topical Solution; Test type: Other — For all analyses, two-tail alpha will be set to 0.05 with no adjustment for multiple comparisons; p = 0.0004, Cochran-Mantel-Haenszel — For all analyses, two-tail alpha will be set to 0.05 with no adjustment for multiple comparisons

ADVERSE EVENTS:
Time Frame: From subject's first study medication application to the end of the study (visit 8), up to 106 days. the end of the subject's last visit. 106.
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a study medication(s) and which does not necessarily have a causal relationship with the study medication. Thus any new, clinically relevant worsening of an existing sign, symptom or disease, should be considered an AE.
Arm/Group | A-101 Vehicle | A-101 (32.5%) Topical Solution | A-101 (40%) Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/57 | 2/57
Other Adverse Events (participants affected / at risk) | 15/58 | 9/57 | 17/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A-101 Vehicle (N=58) | A-101 (32.5%) Topical Solution (N=57) | A-101 (40%) Topical Solution (N=57)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — Invasive ductal carcinoma
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 — right leg laceration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A-101 Vehicle (N=58) | A-101 (32.5%) Topical Solution (N=57) | A-101 (40%) Topical Solution (N=57)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Axillary Pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 2 | 0
Rhinitis allergic (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 1
Tinea Cruris (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2
Viral upper respiratory infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood glucose increase (Investigations) | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 1
Oedema Peripheral (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Insomnia (Nervous system disorders) | 0 | 0 | 1
Dementia (Psychiatric disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Blepharitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Contusion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acrochordon excision (Surgical and medical procedures) | 0 | 0 | 1
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0
Injection (Surgical and medical procedures) | 0 | 0 | 1
Skin neoplasm excision (Surgical and medical procedures) | 0 | 0 | 1
Migraine (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and investigators agree to not publish the results of this study without the permission of the sponsor.